CLINICAL TRIAL: NCT04565964
Title: Association Between Household Health Behaviors and Asthma in Children
Acronym: ABHHBaAiC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202006172RIND
Record Dates: First submitted 2020-09-03; First posted 2020-09-28 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-09

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health behaviors (Other): Health behavior intervention for one month will be provided to every participant. We will teach children's guardians (care-giver) how to change the health behaviors to clean indoor environment, including the health behaviors in bedroom, kitchen room, restroom, refrigerator, washing machine, and incense burning hall.
  Interventions: Other: change the health behaviors to clean indoor environment

INTERVENTIONS:
Other: change the health behaviors to clean indoor environment — Sheets and all covers should be wash weekly. Clean indoor environment with a vacuum cleaner twice a week

SUMMARY:
This study plan to study the association between household health behavior (cleaning habits) and children's asthma. In addition, reconfirm the health effects of indoor environmental exposure to phthalates plasticizers, mite, fungi, and bacteria, and cockroaches on children's asthma. Thus, the investigators can provide a non-pharmacological intervention to reduce the disease burden of children's asthma and allergic diseases.

DETAILED DESCRIPTION:
The investigators plan to invite 80 children, aged 7-12 years-old who have physician-diagnosed asthma, and another age- and gender-matched children without asthma to join our study. First, obtaining clinical data of disease status, and ask participants to fill out questionnaires after recruiting. Second, participants have to record body temperature, peak expiratory flow, heart rate, finger O2 saturation percentage, asthma attack frequency continuously by care-giver every day. Third, the investigators will perform indoor environmental assessments in the subject's house, including indoor air quality, dust samples, culture for fungi and bacteria, and cockroaches. The investigators will also count the dust mites and measure phthalates concentration in every dust sample.

Then, health behavior intervention for one month will be provided to every participant. The investigators will teach children's guardians (care-giver) how to change the health behaviors to clean indoor environment, including the health behaviors in bedroom, kitchen room, restroom, refrigerator, washing machine, and incense burning hall. After 1 months, the investigators will investigate whether changing health behavior affects the exposure of phthalates, dust mites, fungi, bacteria, and cockroaches, and evaluate the effects of health behavior intervention on the clinical status of children's asthma. Children's asthma severity assessment will be recorded by ACT and also by symptomatology every day. Household health behaviors (cleaning habits) questionnaires also will be completed per week and continuously for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 7-12 years-old who have physician-diagnosed asthma
* stable patient

Exclusion Criteria:

* acute allergies
* severe brain and heart disease
* mental illness

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2020-12-29 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Peak expiratory flow changes | one month
  Using peak flow meter to monitor the participant's peak expiratory flow values in the morning and evening to effectively evaluate subject's asthma status.
fractional concentration of exhaled nitric oxide | one month
  Before and after the intervention, test for the levels of fractional exhaled nitric oxide in the hospital to evaluate the condition of airway inflammation.
Pulmonary function test (FVC) | one month
  Before and after the intervention, test for the volumes of the forced vital capacity (FVC) in the hospital as an indicator of asthma status.
Pulmonary function test (FEV1) | one month
  Before and after the intervention, test for the volumes of the forced expiratory volume in one second (FEV1) in the hospital as an indicator of asthma status.
Pulmonary function test (FEV1/FVC ratio) | one month
  Before and after the intervention, test for the FEV1/FVC ratio in the hospital as an indicator of asthma status.
Symptomatology (cough) | one month
  Asthma symptom is recorded daily by caregivers.
Symptomatology (wheezing) | one month
  Asthma symptom is recorded daily by caregivers.
Symptomatology (chest tightness) | one month
  Asthma symptom is recorded daily by caregivers.
dust mites allergen concentrations | one month
  Before and after the intervention, allergen concentrations will be sampled in a fixed area in the subject's bedroom, and dust mites' antibody will be analyzed in the laboratory.
phthalates concentrations | one month
  Sampling in a fixed area in the subject's bedroom, and phthalates concentration will be analyzed in the laboratory.
cockroach numbers | one month
  Before and after the intervention, count the numbers of cockroach will be sampled for every week, in a fixed area in the subject's bedroom.

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Chen Su, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Chung-Shan, Taiwan

IPD SHARING:
Plan to Share IPD: No